CLINICAL TRIAL: NCT06380790
Title: Effect of Laser-aided Circumferential Supracrestal Fiberotomy on the Rate of Leveling and Alignment of Mandibular Anterior Crowding: A Randomized Controlled Clinical Trial
Brief Title: Effect of Laser-aided Csf on the Rate of Leveling and Alignment of Mandibular Anterior Crowding
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sarah Khaled Mohamed Hamed Abdelkader, Orthodontic resident, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 8423
Record Dates: First submitted 2024-03-24; First posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Orthodontics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Other): Placebo laser-aided csf
  Interventions: Other: placebo laser-aided csf
- Intervention (Other): Laser-aided csf before leveling and alignment
  Interventions: Procedure: Laser-aided csf

INTERVENTIONS:
Procedure: Laser-aided csf — Laser-aided csf before leveling and alignment
  Arms: Intervention
Other: placebo laser-aided csf — placebo laser-aided csf before leveling and alignment
  Arms: Control

SUMMARY:
To test the effect of laser-aided circumferential supracrestal fiberotomy on the rate of leveling and alignment

ELIGIBILITY:
Inclusion Criteria:

* Patients indicated for orthodontic treatment 18-25 years
* full permanent dentition (not necessarily third molars)
* mandibular anterior crowding
* no visible anomaly of enamel
* good oral hygiene

Exclusion Criteria:

* patients with mandibular anterior teeth with advanced caries, prosthetic restorations or dental anomalies
* patients with dentofacial deformities or medical problems
* patients indicated for extractions as a part of orthodontic treatment
* patients with severe mandibular gingival inflammation/periodontitis
* pregnant female patients
* patients with previous orthodontic treatment
* patients with previous mandibular extractions except third molars
* patients taking medications that could alter orthodontic treatment
* patients with clefts,syndromes, systemic diseases

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Rate of tooth movement | 4 months
  Rate of leveling and alignment of mandibular incisors

SECONDARY OUTCOMES:
Pain level | 1 week
  Visual Analogue Scale
Periodontal health | 4 months
  Gingival index

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry cairo university, Cairo, Egypt